CLINICAL TRIAL: NCT04076800
Title: Comparison of the Effects of a Standardized Acupuncture Treatment and Sham Acupuncture on Insulin Doses in Insulin-treated Patients With Type 2 Diabetes. A Randomized, Single-blind, Crossover Study.
Brief Title: Acupuncture and Insulin Doses in Insulin-treated Type 2 Diabetes
Acronym: ACUDIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13181
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: acupuncture; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatment will include use of somatic points (SP6; ST36; KI3; CV4; CV12; TE5; LI4; LI11; YinTang; ST28; BL23; BL22; BL20; BL13) and auricular points (most tender point on palpation with pressure feelers of 400 gr on Stomach, Endocrine, Spleen, Kidney, Hungry, Shen man and Pancreas auricular points).

SUMMARY:
This study is a randomized, single blinded, cross-over interventional study for evaluating the effect of acupuncture versus sham acupuncture in diabetic type 2 patient in insulin treatment. Primary end-point of the study is the difference of daily units of insulin between treatment and control group; secondary end point are the variation of glycated hemoglobin levels, lipids panel (total cholesterol, low density lipoprotein, high density lipoprotein, triglycerides), C reactive protein and adiponectin. Variation of epicardial fat thickness will be also evaluated by echography. Acupuncture and sham treatment will be administered twice a week for 3 months and, after a pause of one month and cross-over between groups for other three months. Acupuncture treatment will include use of somatic points (SP6; ST36; KI3; CV4; CV12; TE5; LI4; LI11; YinTang; ST28; BL23; BL22; BL20; BL13) and auricular points (most tender point on palpation with pressure feelers of 400 g on Stomach, Endocrine, Spleen, Kidney, Hungry, Shen man and Pancreas auricular points). Sham acupuncture will be applied distal from acupuncture points and areas used for treatment, with shallow insertion and without manipulation of the needle (15 needles in total on thorax, abdomen, back, arms and legs).

ELIGIBILITY:
Inclusion Criteria:

* type 2 Diabetes Mellitus
* insulin therapy > 20 UI daily for at least 6 months
* HbA1c < 69 mmol/mol

Exclusion Criteria:

* Class I Psychiatric illness not adequately treated
* Actual pregnancy or breastfeeding, or pregnancy planning.
* Corticosteroid treatment
* Severe heart failure (NYHA III-IV)
* Severe renal failure (pre-dialysis o dialysis),
* Severe liver insufficiency (overt cirrhosis)
* Severe respiratory failure (oxygen therapy)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Insulin daily doses | 12 weeks
  Doses of insulin after standardized titration

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  Variations of HbA1c from beginning to end of each treatment phase

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetologia AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No